CLINICAL TRIAL: NCT06389526
Title: A Phase 1, Multicenter, Open-Label Study of CHS-1000 as a Single Agent and in Combination With Toripalimab-tpzi in Participants With Advanced or Metastatic Solid Tumors
Brief Title: A Study of CHS-1000 in Participants With Advanced or Metastatic Solid Tumors
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Coherus Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CHS-1000-01
Record Dates: First submitted 2024-04-25; First posted 2024-04-29 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Advanced or Metastatic Solid Tumors
Keywords: CHS-1000; Tumors; Toripalimab; ILT4; LILRB2
MeSH Terms: conditions — Neoplasms | interventions — toripalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part A: Single Agent CHS-1000 (Experimental)
  Interventions: Biological: CHS-1000
- Part B: Combination Agents CHS-1000 + Toripalimab (Experimental)
  Interventions: Biological: CHS-1000; Biological: Toripalimab

INTERVENTIONS:
Biological: CHS-1000 — Specified dose on specified days
Biological: Toripalimab — Specified dose on specified days
  Other Names: Loqtorzi; Toripalimab-tpzi
  Arms: Part B: Combination Agents CHS-1000 + Toripalimab

SUMMARY:
The primary purpose of this trial is to assess the tolerability and safety of CHS-1000 alone and in combination with toripalimab-tpzi in participants with advanced solid tumors.

ELIGIBILITY:
Key Inclusion Criteria:

* Histopathologically or cytologically confirmed diagnosis of advanced or metastatic unresectable solid tumors (excluding glioblastoma multiforme (GBM)) by tissue biopsy or archival tumor specimen. Unresectable tumors are defined as tumors with lesions in which clear surgical excision margins cannot be obtained, in close proximity to major blood vessels, not with oligometastatic and with advanced organ and lymph node (LN) involvement, and not leading to significant functional compromise as determined by surgical consult or Tumor Board.
* Participants must have been previously treated or be ineligible for, or intolerant of, available approved standard therapies known to confer clinical benefit (including immunotherapy), or for whom no effective standard therapy exists.
* At least 1 measurable lesion based on Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 as determined by the investigator.

Key Exclusion Criteria:

* Concurrent enrollment in another clinical study or participation in another clinical study within 28 days prior to the 1st dose of CHS-1000, except for observational (noninterventional) studies or the follow-up period of an interventional study.
* Current or prior use of systemic anticancer treatment, including but not limited to chemotherapy, immunotherapy, biologic treatment, hormone therapy, and targeted therapy, if within 8 weeks or 5 half-lives (whichever is shorter) for biologic therapies, or if within 28 days for most other anticancer therapies, prior to the 1st dose of CHS-1000.
* Concurrent or prior radiotherapy within 28 days prior to the 1st dose of CHS-1000 or unresolved treatment-related radiation toxicity. Limited local radiotherapy for palliative intent (eg, to a single site of metastatic disease) is permitted within 28 days prior to the 1st dose of CHS-1000 provided that the participant has no evidence of or has recovered from any treatment-related radiation toxicity.

Note: Other protocol-defined inclusion and exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-02-15 (Estimated); Primary Completion 2028-05-30 (Estimated); Study Completion 2028-05-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Treatment-Emergent Adverse Events (TEAEs) | Up to approximately 27 months

SECONDARY OUTCOMES:
Maximum Observed Concentration (Cmax) | Up to approximately 27 months
Area Under the Concentration-time Curve (AUC) | Up to approximately 27 months
Terminal Half-life (t1/2) | Up to approximately 27 months
Number of Participants with Antidrug Antibodies | Up to approximately 27 months
Investigator-assessed Objective Response Rate (ORR) | Up to approximately 27 months
Duration of Response (DoR) | Up to approximately 27 months
Disease Control Rate (DCR) | Up to approximately 27 months
Time to Response (TTP) | Up to approximately 27 months
Progression-free Survival (PFS) | Up to approximately 27 months
Landmark PFS Rate | Month 6, Month 12

IPD SHARING:
Plan to Share IPD: No